CLINICAL TRIAL: NCT02331667
Title: The Effect of Diet on Learning Abilities for Children in Kindergarden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Collaborators: NORCE Norwegian Research Centre AS (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Jannike Øyen, PhD, Scientist, National Institute of Nutrition and Seafood Research, Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014/1396
Record Dates: First submitted 2014-12-17; First posted 2015-01-06 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Performance
Keywords: Diet; Vitamin-D; Meat; Fatty fish; Iodine; fatty acid; Intervention study; Wechsler Preschool and Primary Scale of Intelligence; Strengths and Difficulties Questionnaire; Nine hole peg test
MeSH Terms: interventions — Seafood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seafood (Experimental): Intervention with meals consisting of seafood (herring and mackrell).
  Interventions: Other: Seafood
- Non-seafood (Experimental): Intervention with meals constisting of non-seafood (meat).
  Interventions: Other: Non-seafood

INTERVENTIONS:
Other: Seafood — The aim is to investigate the effect of meals consisting of mackrel and herring on learning abilities by using a two-armed individually randomized non-blinded intervention trial.
  Arms: Seafood
Other: Non-seafood — The aim is to investigate the effect of meals consisting of meat on learning abilities by using a two-armed individually randomized non-blinded intervention trial.
  Arms: Non-seafood

SUMMARY:
The main aim of this intervention study is to test the effect of diet on improvement in cognitive performanc in kindergarden children aged 4-6 years. Children will be randomly allocated into two groups, one consuming prepared meals with herring or mackerel for four months, and one group consuming meals containing meat as a control group.

DETAILED DESCRIPTION:
Positive effects of n-3 long chain polyunsaturated fatty acids (PUFAs), as provided by fatty fish intake, on cognitive functions are widely accepted, but so far there is no clear evidence from randomized intervention studies in children and young adults, although fish intake has been positively associated with cognitive functions in observational studies. The main aim of this study is to test the effect of diet on improvement in cognitive performance in kindergarden children aged 4-6 years. In the intervention study, children will be randomly allocated into two groups, one consuming prepared meals with herring or mackerel for four months, and one group consuming meals containing meat as a control group. The children (n=200) will consume the prepared meals three times a week. Cognitive performance of the children will be tested at study start and end using the the Wechsler Preschool and Primary Scale of Intelligence (WPPSI_III) and nine hole peg test. Children will be screened for mental health problems in the Strengths and Difficulties Questionnaire (SDQ), which is a global measure of children's mental health. Compliance will be monitored by documentation of study fish intake and measuring fatty acid status. For a more detailed investigation of effects of increased herring and mackerel intake, before and after intervention blood and urine will be collected for lipidomic analysis (metabolites), vitamin D and iodine determination and genotyping (fatty acid metabolism and inflammation).

ELIGIBILITY:
Inclusion Criteria:

* Being 4-6 years old.
* Sufficient command of the Norwegian language of child to participate in cognitive testing and of child and parents to comply with study requirements according to investigators estimation.

Exclusion Criteria:

* Known food allergies

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 233 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
WPSSI-III and Nine Hole peg test. | 5 months
  The intervention study aims to test the effect of diet on improvement in cognitive performance measured by WPPSSI-III and Nine Hope Peg test in kindergarten children.

SECONDARY OUTCOMES:
Mercury | 5 months
  Total hair mercury concentration
Mental health | 5 months
  Strengths and difficulties questionnaire (SDQ)
Sleep | 5 months
  Questionnaire report by parent
B-vitamines | 5 months
  Serum: Cobalamin, Flavin Mononucleotide, Folate, HCC-index, HK:XA, MMA, N1-methylnicotinamide, PA, PL, PLP, Riboflavin, tHcy, Thiamin, Thiamin monophosphate
Cholline pathway | 5 months
  Serum: Betaine, Choline, Dimethylglycine, Glycine, Serine, TMAO
Tryptophan pathway | 5 months
  Serum: 3-Hydroxyanthranilic acids, 3-Hydroxykynurenine, Anthranilic acid, Kynurenic acid, Kynurenine, Tryptophan, Xanthurenic acid, Nicotinamide, Picolinic acid, Quinolic acid c acid,
Amino acids | 5 months
  Serum: 1-MH, 3-MH, ADMa, Alanine, Arginine, Asparagine, Aspartic acid, Cystathionine, Glutamic acid, Glutamine, Histidine, Homoarginine, Isoleucine, Leucine, Lysine, Methionine, Methionine sulfoxide, Ornithine, Phenylalanine, Proline, SDMA, Threonine, Total Cysteine, Trimethyllysine, Tyrosine, Valine
Inflammation | 5 months
  Serum: Kynureine/Tryptophan-ratio, Neopterin, PAr index
Creatinine | 5 months
  Serum Creatinine
Fatty acids | 5 months
  RBC: C16:3n3 (HTA), C20:5n3 (EPA), C22:6n3 (DHA), Sum n-3, C18:2n6 (LA), C30:3n6 (ETE), C20:4n6 (AA), C22:4n& (AdA), Sum n-6, Ratio n-3/n-6, C14:0, C16:0, C18:0, C22:0, C16:1, C18:1, C24:1n9
Ferritin | 5 months
  Serum ferritin
25-hydroxyvitamin D | 5 months
  serum 25(OH)D3
Iodine concentration | 5 months
  Urinary iodine concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Eide Graff, PhD, Study Director — NIFES, Postboks 2029 Nordnes, 5817 Bergen, Norway
Locations (1):
- NIFES, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
The results will be published in international journals.
Supporting Information: Study Protocol
Time Frame: From study start until 2023
Access Criteria: Upon request to the project manager.

REFERENCES:
- [Derived] Solvik BS, Oyen J, Kvestad I, Markhus MW, Ueland PM, McCann A, Strand TA. Biomarkers and Fatty Fish Intake: A Randomized Controlled Trial in Norwegian Preschool Children. J Nutr. 2021 Aug 7;151(8):2134-2141. doi: 10.1093/jn/nxab112. PMID 33978160
- [Derived] Solvik BS, Strand TA, Kvestad I, Markhus MW, Ueland PM, McCann A, Oyen J. Dietary Intake and Biomarkers of Folate and Cobalamin Status in Norwegian Preschool Children: The FINS-KIDS Study. J Nutr. 2020 Jul 1;150(7):1852-1858. doi: 10.1093/jn/nxaa111. PMID 32338756
- [Derived] Oyen J, Kvestad I, Midtbo LK, Graff IE, Hysing M, Stormark KM, Markhus MW, Baste V, Froyland L, Koletzko B, Demmelmair H, Dahl L, Lie O, Kjellevold M. Fatty fish intake and cognitive function: FINS-KIDS, a randomized controlled trial in preschool children. BMC Med. 2018 Mar 12;16(1):41. doi: 10.1186/s12916-018-1020-z. PMID 29530020